

## PARTICIPANT INFORMATION DOCUMENT

#### BRIEF SURVEY OF CORRECTION OFFICERS

## **Key Information**

- This is a research project to better understand knowledge, attitudes, and skills related to a "Targeted Educational Campaign" (TEC) whose aim is to give Correction Officers the information they need to identify young people with possible early psychosis.
- The research study is voluntary. You can decide not to participate or withdraw at any time with no consequences.
- The survey will measure TEC-related knowledge, attitudes, and skills, and should take less than 10 minutes to complete.
- We do not foresee any risks for Correction Officers.

### **Purpose and Overview**

The purpose of this study is to briefly collect data on knowledge, attitudes, and skills related to a "Targeted Educational Campaign" (TEC) being carried out in three jails at Rikers Island. The goal of the TEC is to give Correction Officers the information they need to identify young people with possible early psychosis who are not yet receiving mental health services in the jail, and refer them to Correctional Health Services.

This study is funded by a grant from the National Institute of Mental Health.

### Voluntary

Participation in this survey is your choice. If you decide not to participate, or if you later decide to stop participating, you will not lose any benefits to which you are otherwise entitled. A decision not to participate or to withdraw participation will not affect your employment status. Below you will be given a description of the risks, benefits, and alternatives to participating in the survey. Before you make your decision, please read through this form carefully. Please ask any questions about anything that is not clear.

#### **Procedures**

We are giving this survey to a large group of Correction Officers before the "Targeted Educational Campaign" (TEC) is implemented, and then again at 6-months into the TEC, and at 12-months into the TEC. The survey will measure knowledge, attitudes, and skills, and should take less than 10 minutes to complete.

### **Risks and Inconveniences**

We do not foresee any risks for Correction Officers. Your participation is completely voluntary and the information collected will be confidential and anonymous, and will not be disclosed outside of the research team.

#### **Benefits**

# NYSPI IRB Approved 7771 5/13/2019 -> 4/21/2020

## **Brief Survey of Correction Officers**

There may be no direct benefits to you, but significant potential knowledge will be gained from the research. The research will provide an understanding of the impact of a educational campaign in a jail to improve detection of untreated psychosis among detainees.

# **Confidentiality**

All information collected will be confidential and anonymous and will not be disclosed outside of the research team. We will keep all records private and confidential to the extent permitted by law. Your name and other identifiers will not be included in the notes or dataset and each participant in the study will be assigned a unique ID number.

Surveys will be made anonymous using a unique ID. For example, on the front page of the survey, you will be asked: "What is the first letter of your middle name?" and several other questions so that you can create a unique identification code (such as JB22, TF18) to ensure that you remain anonymous, while allowing us to match any participants who complete a later survey (at 6 months or 12 months). The information collected could be used for future research studies or distributed to another investigator for future research studies, without identifiers.

Records will be made available to Federal, State, and Institutional regulatory personnel if records are reviewed as part of routine audits.

Relevant research results will be made available through publications in scientific journals and presentations to conferences for the mental health research community and corrections community, but will not be directly disclosed to you.

# **Study Compensation**

There is no compensation for this study

#### **Ouestions**

You are encouraged to ask us any questions about the study at any time. You can ask questions before, during, or after the survey. You can also contact the lead researcher, Dr. Michael Compton, at: (646)-774-8476 or mtc2176@cumc.columbia.edu. He will answer to the best of his ability any questions or concerns that you have now or in the future about the research. For any questions about your rights as a research participant, if you want to provide feedback, or if you have a complaint, you may call the New York State Psychiatric Institute (NYSPI) Institutional Review Board (IRB), which is the committee that protects the rights of participants in research studies, at (646)-774-7155 during regular office hours.

### **Consent to Participate in the Survey**

You understand that participation is voluntary, and it is up to you to decide if you want to participate in the survey. Participating involves completing some brief survey questions. If you proceed to the survey on the next page, you are giving your consent to be a participant.